CLINICAL TRIAL: NCT02834234
Title: Genomic Analysis of Peritoneal Mesothelioma by CGH Arrays
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50828
Record Dates: First submitted 2016-04-27; First posted 2016-07-15 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Peritoneal Mesothelioma
Keywords: mesothelioma; peritoneum; genomic; CGH arrays
MeSH Terms: conditions — Mesothelioma | interventions — Comparative Genomic Hybridization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — mesothelioma tumor specimen and normal tissue specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peritoneal mesothelioma specimens: The group harbors only patients who received the diagnosis of peritoneal mesothelioma after surgery. All patients are included in this group.
  The CGH arrays will be realized on frozen samples (for the comparative genomic analysis).
  Interventions: Genetic: comparative genomic analysis

INTERVENTIONS:
Genetic: comparative genomic analysis — DNA and RNA extraction will be performed in Lyon University hospital (genomic platform) using commercially available kit. Percentage of tumors cells will be controlled by stained section before extraction. The CGH arrays will be realized on frozen samples in Lille (genomic platform). Pangenomic Agilent array will be used. Micro-array include 180000 probes. Analysis will be performed in Lille (genomic platform / department of BioInformatics) with Marie Brevet. Data will be processed from the log2 transformed data into normalization with the WACA method. Then copy number variation will then be identified with Circular Binary Segmentation. Copy number variations will be called as gain or deletion according to the log2 ratio distribution and the percent of tumoral cells. Using matched tumoral and normal DNA will eliminate Copy Number Polymorphisms. We will construct non supervised hierarchical analyses to study the classification of peritoneal mesothelioma based on copy number variation

SUMMARY:
Peritoneal mesothelioma is a rare disease representing one third of all mesothelioma and nothing is known about molecular characteristics of this disease. As main cancers, genetic heterogeneity is probable. This genomic profiling associates Comparative Genomic Hybridization (CGH) array, BAP1 sequencing and gene expression in order to discover a biomarker that could be used in the treatment of this rare disease. Corresponding histopathological and immunohistochemical report as all clinical data are available. All data with be merged to underline a few genes of interest on which we will focus our next investigations. Depending of our preliminary results, BAP1 mutations are expected, as it was also described in pleural mesothelioma. Mutations in oncogenic drivers that could be targeted by specific therapy will be on particular interest in management of this rare disease with bad prognosis.

ELIGIBILITY:
Inclusion Criteria:

* surgical biopsy od the peritoneal tumor with frozen samples
* age > 18 years old

Exclusion Criteria:

* absence of peritoneal mesothelioma
* absence of frozen samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of peritoneal mesothelioma
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
BAP1 mutations | Day 0
  CGH Array